CLINICAL TRIAL: NCT00498784
Title: A Multicenter, Open Labelled, Uncontrolled, Phase IV Clinical Study to Evaluate the Health-related Quality of Life and Sexual Well-being in Young (18-35) Healthy Mirena Users Switching From OC, Over the First Year Post-insertion.
Brief Title: HR-QoL and Sexuality in Mirena Inserted Contraception Users
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Medical Affairs Therapeutic Area Head, Bayer Healthcare AG
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 91458; 2005-002955-42 (EudraCT Number); 309663 (Other: Company internal)
Record Dates: First submitted 2007-07-09; First posted 2007-07-10 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Contraception
Keywords: Intra-uterine contraception; Intrauterine Devices
MeSH Terms: interventions — Levonorgestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Mirena

INTERVENTIONS:
Drug: Mirena — Mirena 52mg during 1 year

SUMMARY:
The purpose of this study is to evaluate the changes in the quality of life, as well as in the sexual activity, in women inserted with MIRENA, a hormonal contraceptive intra-uterine system, over the first 12 months of use. Patients switching from oral contraception to an intrauterine contraceptive device (here: MIRENA) will be observed in the first year post MIRENA insertion.

ELIGIBILITY:
Inclusion Criteria:

* Healthy woman willing to, or having to switch from her OC to another contraceptive method

Exclusion Criteria:

- Any contraindication to Mirena insertion/use

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 141 (Actual)
Dates: Start 2005-11; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Health-related QoL score | 1 year

SECONDARY OUTCOMES:
Sexuality Index, treatment satisfaction, usual safety outcomes | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Bordeaux, Gironde, France